CLINICAL TRIAL: NCT02710201
Title: A Randomized-controlled Trial of Social Norm Interventions to Increase Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Merced (Other)
Responsible Party: Principal Investigator, Linda Diane Cameron, Professor of Psychology, University of California, Merced
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: UCM13-00012
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): No feedback on progress of other participants.
- Descriptive Social Norm (Experimental): Average physical activity of other participants in study conveyed to this group.
  Interventions: Behavioral: Descriptive Social Norm
- Descriptive-plus-Injunctive Social Norm (Experimental): Average physical activity of other participants in study and message of approval or disapproval (depending on how one is faring compared to others) conveyed to this group.
  Interventions: Behavioral: Descriptive-plus-Injunctive Social Norm

INTERVENTIONS:
Behavioral: Descriptive Social Norm
  Arms: Descriptive Social Norm
Behavioral: Descriptive-plus-Injunctive Social Norm
  Arms: Descriptive-plus-Injunctive Social Norm

SUMMARY:
Objective: Physical activity confers numerous health benefits, yet few adults meet recommended physical activity guidelines. The impact of brief messages providing feedback on physical activity was tested in this study. Methods: Young adults were randomly assigned to one of three conditions: (1) feedback on how active others were, (2) feedback on how active others were plus a message of approval or disapproval depending on whether the participant was more or less active than average, or (3) no feedback (control condition). Participants used pedometers for eight weekdays and recorded their step counts each evening. The group receiving feedback on how active others were got information about the average number of steps taken by group members the previous day. The group that also received approval or disapproval received feedback about the group average, as well as a sad face if the participant was below the average or a happy face if the participant was above the average. The control group received no feedback throughout the study. Impacts of these feedback messages were compared on number of steps taken during the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older

Exclusion Criteria:

* Answering yes to any questions on the Physical Activity Readiness Questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Number of steps | Two weeks
  Number of steps taken daily, as measured by a pedometer.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wally CM, Cameron LD. A Randomized-Controlled Trial of Social Norm Interventions to Increase Physical Activity. Ann Behav Med. 2017 Oct;51(5):642-651. doi: 10.1007/s12160-017-9887-z. PMID 28213634